CLINICAL TRIAL: NCT04263415
Title: The Effects of Semaglutide on Modulation of Taste Sensitivity, Tongue Tissue Transcriptome, Gastric Emptying and Central Neural Responses in Women With PCOS and Obesity: a Randomized, Single-blind, Placebo-controlled Clinical Trial
Brief Title: The Effects of Semaglutide on Taste, Tongue Tissue Transcriptome, Gastric Emptying and Central Neural Response in Women With PCOS and Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, Clinical professor, Head of the Department of Endocrinology, Diabetes and Metabolic Diseases, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sema in PCOS
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: PCOS; Semaglutide; Taste, Altered; Tongue Tissue Transcriptome; Gastric Emptying; Central Neural Response
MeSH Terms: conditions — Dysgeusia | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: a randomized, single-blind, placebo-controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group P (Placebo Comparator): once-weekly injection with placebo pen.
  Interventions: Other: Placebo
- group S (Experimental): Once-weekly application of semaglutide
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — semaglutide inrun period of 4 weeks with 0.5mg/week s.c. followed by 1mg/week sc for 12 weeks
  Other Names: Ozempic
  Arms: group S
Other: Placebo — once-weekly injection with placebo pen for 16 weeks
  Arms: group P

SUMMARY:
The purpose of the study is to explore the effects of GLP-1 receptor agonist (GLP-1 RA) semaglutide on modulation of taste sensitivity, tongue tissue transcriptome, modulation of neural response in central reward processing regions and gastric emptying rate. In addition, we aim to investigate the associations between semaglutide induced modulation of taste sensitivity, neural responses and gastric emptying with changes in body mass, eating- behavioural pattern, food perception and food intake.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent
* Diagnosed with PCOS by Rotterdam criteria
* BMI > 30 kg/m2
* Age 18 years-menopause

Exclusion Criteria:

* Severe psychiatric disease including schizophrenia, paranoid psychosis, bipolar disorder or mental retardation
* Current history of neurological disease including traumatic brain surgery
* Current history of diagnosis of type I or type II diabetes or plasma haemoglobin A1c 6.5% at inclusion
* Impaired hepatic function (liver transaminases>3 times upper normal limit)
* Impaired renal function (estimated glomerular filtration rate (eGFR)< 50 ml/min
* Impaired pancreatic function (any history of acute or chronic pancreatitis and/or amylase >2 times upper limit)
* Bleeding disorders
* Women who are pregnant, breast feeding or have intention of becoming pregnant within the next 9 months
* Women who are planning any operation within the next 6 months
* History of medullary thyroid carcinoma (MTC) and/or family history with MTC and/or multiple endocrine neoplasia syndrome type 2
* Cardiac problems defined as decompensated heart failure (New York Herat Association functional class III or IV), unstable angina pectoris, and/or myocardial infarction within the last 12 months
* Uncontrolled hypertension (systolic blood pressure > 180 mmHg, diastolic blood pressure > 110 mmHg
* Receiving GLP-1 agonist within the last 12 months
* Use of any weight-lowering pharmacotherapy within the preceding 3 months
* Contraindication for MR scanning (magnetic implants, pacemaker, claustrophobia etc)
* Any condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
to investigate the effect of semaglutide on taste perception as change in taste sensitivity detected by chemical gustometry evaluated with "Taste strips" test | Changes in taste perception from baseline up to the end of 12th week.
CO-PRIMARY END-POINT : to investigate alteration of transcriptomic profile of human tongue tissue as changes in expression level from baseline to follow up after 12 weeks of treatment, measured by RNA sequencing | Change in transcriptomic profile from baseline up to the end of 12th week.

SECONDARY OUTCOMES:
Change in neural response to visual food cues and taste task as assessed by functional MRI | Change in neural response to visual food cues and taste task from baseline up to the end of 12th week.
Change in eating behaviour by using a Slovenian translation of Three-Factor Eating Questionnaire TFEQ-R18. | Change in eating behaviour from baseline to the end of 12th week of therapy.
Change in body weight measured with body weight scale to the nearest 1 kg | Change in body weight from baseline to the end of 12th week of therapy.
Change in body fat mass assessed by a Dual Energy X-ray Absorptiometry | Change in body fat mass from baseline to the end of 12th week of therapy.
The impact of sema on gastric emptying | Change of gastric emptying from baseline to the end of 12th week of therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensterle M, Ferjan S, Battelino T, Kovac J, Battelino S, Suput D, Vovk A, Janez A. Does intervention with GLP-1 receptor agonist semaglutide modulate perception of sweet taste in women with obesity: study protocol of a randomized, single-blinded, placebo-controlled clinical trial. Trials. 2021 Jul 19;22(1):464. doi: 10.1186/s13063-021-05442-y. PMID 34281590